CLINICAL TRIAL: NCT06330298
Title: Improving Social Cognition and Social Behaviour in Various Brain Disorders.
Acronym: T-ScEmo4ALL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202000479
Record Dates: First submitted 2023-12-12; First posted 2024-03-26 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Stroke; Multiple Sclerosis; Brain Tumor
Keywords: Neuropsychology; Treatment; Social cognitive disorders; Emotion recognition; Theory of Mind; Social behaviour; Neurological disorders; Stroke; Brain tumour; Mulitple Sclerosis
MeSH Terms: conditions — Stroke; Multiple Sclerosis; Brain Neoplasms; Social Behavior; Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: Experimental condition T0, baseline measurement at point of inclusion (at least > 6 months post-acute injuries) T1, post measurement within 2 weeks after treatment T2, follow-up measurement within 3 - 5 months after treatment
  Waiting list condition T0, baseline measurement at point of inclusion (at least > 6 months post-acute injuries) T1, post measurement within 3 months after T0 T2, follow-up measurement within 3 - 5 months after T1
  TBI group T1, post measurement within 2 weeks after treatment T2, follow-up measurement within 3 - 5 months after treatment
  The participating patients are randomly allocated into two groups: an experimental condition and a waiting list condition.
  In addition, a group of patients with Traumatic Brain Injury will receive T-ScEmo following regular care.
Who Masked: Investigator
Masking Description: The neuropsychologist who leads T1 and T2 measurements will be masked for the fact of which patient will be draw in which clinical condition (experimental group or control group), however this cannot be guaranteed since patients may talk about their experience.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental condition: Receives T-ScEmo Treatment (Experimental): Experimental group. Receives T-ScEmo Treatment during the study between T0 and T1
  Interventions: Behavioral: Treatment social cognition and emotion regulation (T-ScEmo)
- Waiting list group: Will be on waiting list instead of treatment (No Intervention): Waiting list group: Will be on waiting list for instead of the treatment for the duration of the treatment between T0 and T1.

INTERVENTIONS:
Behavioral: Treatment social cognition and emotion regulation (T-ScEmo) — T-ScEmo is a multifaceted treatment protocol that has the overall aim to improve social cognition, regulation of social behaviour and social participation in everyday life (Westerhof et al., 2017; 2019). The treatment includes, in addition to practicing social cognitive skills throughout the treatment, close involvement of a significant other, and homework assignments. The treatment consists of three modules that address 1) perception of social information including facial expressions of emotions, 2) perspective taking and understanding of social information and 3) regulation of social behaviour. The treatment contains 15-one hour live treatment sessions with a neuropsychologist and 5 online practice sessions, once or twice a week. In the online sessions, the patient can practice the information at home as a neuropsychologist is available for questions. When patients find it too difficult to practice individually at home, there is a opportunity to offer these sessions as live sessions
  Arms: Experimental condition: Receives T-ScEmo Treatment

SUMMARY:
Impairments in aspects of social cognition are disorder-transcending: these have been demonstrated in various neurological disorders, such as traumatic brain injury (TBI), stroke, brain tumours (both low grade glioma's and meningioma's) and multiple sclerosis (MS). Social cognition involves processing of social information, in particular the abilities to perceive social signals, understand others and respond appropriately (Adolphs 2001). Crucial aspects of social cognition are the recognition of facial expressions of emotions, perspective taking (also referred to as mentalizing or Theory of Mind), and empathy. Impairments in social cognition can have a large negative impact on self-care, communication, social and professional functioning, and thus on quality of life of patients.

Recently, a first multi-faceted treatment for social cognitive impairments in TBI was developed and evaluated; T-ScEmo (Training Social Cognition and Emotion). T-ScEmo turned out to be effective in reducing social cognitive symptoms and improving daily life social functioning in this particular group, with effects lasting over time (Westerhof-Evers et al, 2017, 2019).

Unfortunately, up till now there are no evidence based, transdiagnostic treatment possibilities available for these impeding social cognition impairments in neurological patient groups, other than TBI. Therefore the aim of the present study is to investigate whether T-ScEmo is effective for social cognition disorders in patients with different neurological impairments, such as stroke (including subarachnoidal haemorrhage (SAH)), brain tumours, MS, infection (meningitis, encephalitis) and other. The secondary objective is to determine which patient related factors are of influence on treatment effectiveness. In short, hopefully this study can contribute to a treatment possibility for social cognition disorders for all patients with various neurological disorders.

It is expected that T-ScEmo will be effective for various neurological disorders, based on previous research of Westerhof-Evers et al. (2017, 2019). Since social cognition disorders within patients with traumatic brain injury do all have the same ethiology it is expected that the treatment will show the same effects for patients with various neurological disorders. Therefore it is expected that patients will improve on social cognition, social participation and quality of life and social behaviour, that these results will last over time.

ELIGIBILITY:
Inclusion Criteria:

* Patients should have social cognitive disorders that show by means of problems in emotion recognition, perspective taking, ToM, showing empathy, or behaviour.
* Patients should have a neurological disorder; stroke (including patients with subarachnoid haemorrhage), Multiple sclerosis (MS), both relapsing remitting, primary and secondary progressive variants, Brain tumours (meningioma's, low grade gliomas) and other categories of neurological disorders including brain damage: (i.e. infections (meningitis, encephalitis), post anoxic encephalopathy, adult survivors of childhood brain tumours).
* Patients should be aged between 18 and 75
* Patients should be in the chronic stage (> 6 months post-acute injuries) or their medical condition should be relatively stable (for patients with a slow progressive conditions), to be judged by the treating medical or psychological specialist, in order to be able to profit from treatment for a reasonable time period.

Exclusion Criteria:

* Serious neurodegenerative or psychiatric conditions (including addiction) interfering with treatment
* Incapacity to act, to be judged by the neuropsychologist and/or neurologist
* Serious cognitive problems (aphasia, neglect, amnesia, dementia) and/or serious behavioural problems (aggression, apathy) interfering with treatment, to be judged by neuropsychologist.
* Serious (other) medical conditions or physical inability hindering patients to come to the hospital/rehabilitation centre
* Not being available of a close other (life partner, family member, close friend) who can fill out the proxy questionnaires
* Not willing to give permission to send important/unexpected findings to the general practitioner.
* Unexpected progression of disease during the study can be a reason to exclude the patient
* Not sufficient command of the Dutch Language.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2021-05-31 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in social behaviour examined by proxy | Through study completion, an average of 8 to 10 months
  The main study parameter will be the difference between baseline (T0) and follow-up (T2) on Dysexecutive Questionnaire Social scales proxy version (DEX-Socproxy; Spikman et al., 2013; Westerhof-Evers, 2017). This scale is scored by the involved proxy of the patient (life partner, family member, friend) and measures the social aspects in daily life: 1) social convention, 2) behavioural-emotional selfregulation 3) metacognition. A higher outcome means more behavioural complaints.

SECONDARY OUTCOMES:
Social cognition: Emotion recognition as assessed using the Eckman-60 faces test | Through study completion, an average of 8 to 10 months
  Performance on neuropsychological test measuring emotion recognition; Eckman-60 faces test (EFT). This test has a range between 0 and 60. A higher outcome means a better performance.
Social cognition: Theory of Mind as assessed using the Happé cartoons test | Through study completion, an average of 8 to 10 months
  Performance on neuropsychological test measuring Theory of Mind; Happé cartoons test. This test has a range between 0 and 36. A higher outcome means a better performance.
Social cognition: Theory of Mind as assessed using the Faux Pas test | Through study completion, an average of 8 to 10 months
  Performance on neuropsychological test measuring Theory of Mind: Faux Pas test. This test has a range between 0 and 10. A higher outcome means a better performance.
Social cognition: assessed using the Hailing Sentence Completion Test | Through study completion, an average of 8 to 10 months
  Performance on neuropsychological test measuring inhibition; Hailing Sentence Completion Test. This test has a range between 1 and 10. A higher outcome means a better performance.
Demographic information | Through study completion, an average of 8 to 10 months
  Demographic information such as age, sex, educational level, will be obtained from medical records and anamnesis.
Self-rated social behaviour as assessed using the Dysexecutive questionnaire Social Scales. | Through study completion, an average of 8 to 10 months
  Self-reated social behaviour will be measured with a self rating on the Dysexecutive questionnaire Social Scales. Measuring the social aspects in daily life: 1) social convention, 2) behavioural-emotional selfregulation 3) metacognition. This scale has a range between 0 and 80. A higher outcome means more complaints.
Self-rated social behaviour as assessed using the Interpersonal Reactivity Index | Through study completion, an average of 8 to 10 months
  Self-rated social behavior will be measured with the Interpersonal Reactivity Index (IRI). This scale has a range between 0 and 108. A higher outcome means less behavioural complaints.
Self-rated social behaviour as assessed using The Dutch version of the BAFQ social scales | Through study completion, an average of 8 to 10 months
  Self-rated social behavior will be measured with The Dutch version of the BAFQ social scales (BAFQ-SOC). Moreover, patients answer if they have changed on that certain topic after brain damage. A higher outcome means less behavioural complaints and more change.
Proxy-rated social behaviour as assessed using the Interpersonal Reactivity Index | Through study completion, an average of 8 to 10 months
  Proxy-rated social behavior will be measured with the Interpersonal Reactivity Index, proxy version (IRI). This scale has a range between 0 and 108. A higher outcome means less behavioural complaints.
Proxy-rated social behaviour as assessed using the Socioemotional Dysfunction Scale | Through study completion, an average of 8 to 10 months
  Proxy-rated social behavior will be measured with the Socioemotional Dysfunction Scale (SDS). This scale has a range between 40 and 200. A higher outcome means more complaints.
Proxy-rated social behaviour as assessed using the Dutch version of the BAFQ social scales | Through study completion, an average of 8 to 10 months
  Proxy-rated social behavior will be measured with the Dutch version of the BAFQ social scales, proxy version (BAFQ-SOC). Moreover, proxies answer if patients have changed on that certain topic after brain damage. A higher outcome means less behavioural complaints and more change.
Alexithymia | Through study completion, an average of 8 to 10 months
  The presence of alexithymia will be measured with a self-rating on the Toronto Alexithymia Scale (TAS-20). This scale has a range between 20 and 100. A higher outcome means more complaints.
Life satisfaction | Through study completion, an average of 8 to 10 months
  Quality of life will be determined with a self-rating on the Life Satisfaction Questionnaire (LSQ-9). This scale has a range between 6 and 54. A higher outcome means a higher subjective quality of life.
(Social) participation as assessed using the Utrecht Scale for Evaluation of Rehabilitation | Through study completion, an average of 8 to 10 months
  The level of societal participation will be measured with the scores on the Utrecht Scale for Evaluation of Rehabilitation (USER-P). A higher outcome means higher participation rate.
(Social) participation as assessed using the Impact on Participation and Autonomy scale | Through study completion, an average of 8 to 10 months
  The level of societal participation will be measured with the Impact on Participation and Autonomy (IPA). A higher outcome means lower participation rate.
Mood and anxiety | Through study completion, an average of 8 to 10 months
  The level of mood and anxiety will be obtained with the Hospital Anxiety and Depression Scale (HADS). This scale has a range between 0 and 42. A higher outcome means more complaints.
Caregiving burden | Through study completion, an average of 8 to 10 months
  The extend to which proxies experience a burden in taking care of the patient wil be measured with the Zarit burden interview. This scale has a range between 0 and 48. A higher outcome means more burden.
Goal attainment | Through study completion, an average of 8 to 10 months
  The extent to which patients in the treatment condition improve on their set treatment goals will be measured with the Goal Attainment Scale (GAS). This scale has a range between 1 and 10. A higher outcome means better attainment.

OTHER OUTCOMES:
Executive functioning as assessed using the Controlled Oral Word Association Test | Baseline
  Only at baseline (T0), the following additional measures will be determined, allowing to control for factors that may interfere with treatment effects.
  Executive functioning will be measured with the Controlled Oral Word Association Test (COWAT).
Executive functioning assessed using the Key Search Test | Baseline
  Only at baseline (T0), the following additional measures will be determined, allowing to control for factors that may interfere with treatment effects.
  Executive functioning will be measured with the Key Search Test of the Behavioural Assessment of the Dysexecutive Syndrome.
Verbal memory | Baseline
  Only at baseline (T0), the following additional measures will be determined, allowing to control for factors that may interfere with treatment effects.
  Verbal memory will be measured with Dutch version of the Rey Auditory Verbal Learning Test (15 Words Test).
Working memory | Baseline
  Only at baseline (T0), the following additional measures will be determined, allowing to control for factors that may interfere with treatment effects.
  Working memory will be measured with the Digit Span Test of the Wechsler Adult Intelligence Scale IV.
Language | Baseline
  Only at baseline (T0), the following additional measures will be determined, allowing to control for factors that may interfere with treatment effects.
  Language will be measured with the semantic fluency test.
Mental speed and attention as assessed using the Trail Making Test | Baseline
  Only at baseline (T0), the following additional measures will be determined, allowing to control for factors that may interfere with treatment effects.
  Mental speed and attention will be measured with the Trail Making Test (TMT).
Mental speed and attention as assessed using the Symbol Digit Modalities Test | Baseline
  Only at baseline (T0), the following additional measures will be determined, allowing to control for factors that may interfere with treatment effects.
  Mental speed will be measured with the Symbol Digit Modalities Test (SDMT).
Premorbid intelligence | Baseline
  Only at baseline (T0), the following additional measures will be determined, allowing to control for factors that may interfere with treatment effects.
  Premorbid intelligence will be measured with Dutch version of the Adult Reading Test (NLV).
Fatigue | Baseline
  Only at baseline (T0), the following additional measures will be determined, allowing to control for factors that may interfere with treatment effects.
  The level of physical and mental fatigue will be measured with the Dutch Multifactor Fatigue Scale (DMFS).
  This scale has a range between 38 and 190. A higher outcome means more complaints.
Health limitations | Baseline
  Only at baseline (T0), the following additional measures will be determined, allowing to control for factors that may interfere with treatment effects.
  Health related physical and practical limitations will be measured with the RAND-36 Health Survey.
  A higher outcome means better functioning.
Coping | Baseline
  Only at baseline (T0), the following additional measures will be determined, allowing to control for factors that may interfere with treatment effects.
  Coping will be measured with the Utrecht Coping List (UCL)
  A higher outcome means a better fitting coping style.

CONTACTS AND LOCATIONS:
Overall Officials: J.M. Spikman, Prof. Dr., Principal Investigator — Department of Neurology - Unit Neuropsychology of the University Medical Center Groningen (UMCG)
Locations (2):
- Netherlands (2):
  - Deventer Hospital, Deventer, Overijssel
  - University Medical Center Groningen, Groningen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Heegers A, Rakers SE, van Twillert S, Moulaert VRM, Gerritsen MMJ, van der Naalt J, Spikman JM, Westerhof-Evers HJ. Social Cognitive Treatment (T-ScEmo) for Various Neurological Patient Groups: Study Rationale and Protocol for a Randomized Control Trial (T-ScEmo4ALL). BMC Neurol. 2025 Mar 27;25(1):129. doi: 10.1186/s12883-025-04125-4. PMID 40148852